CLINICAL TRIAL: NCT04838587
Title: An Epidemiological Surveillance Study to Determine the Incidence of ETEC in Children and Infants in Lusaka.
Acronym: ETEC-Surv
Status: Completed | Type: Observational
Sponsor: Centre for Infectious Disease Research in Zambia (Other)
Collaborators: European and Developing Countries Clinical Trials Partnership (EDCTP) (Other Government); Scandinavian Biopharma AB (Industry); Göteborg University (Other)
Responsible Party: Sponsor
Other Study IDs: 1091-2020
Record Dates: First submitted 2021-02-05; First posted 2021-04-09 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Diarrhea Toddlers; Escherichia Coli Diarrhea
Keywords: Incidence; Epidemiology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — faecal specimen
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 6750 Children <3 years ( 5 sites): A total of 6750 children from the will be identified from the respective health facility catchment area during the Census stage of the study. Each of the 5 health facilities will identify 1350 children under 3 years of age in their respective catchment area. During the Surveillance stage, the participants will be enrolled into the study if and when they present with diarrhoea at the Health facility.
  Interventions: Other: No intervention will be done

INTERVENTIONS:
Other: No intervention will be done — No intervention,Only passive surveillance of Diarrhoea cases will be done

SUMMARY:
Diarrhoea is the one of the top five leading causes of death among children below the age of five years, globally. It is estimated that one in ten deaths in children under five is attributed to diarrhoea. Enterotoxigenic E.coli (ETEC) is one of the major causative agents of moderate-to-severe (MSD) diarrhoea among children both globally and in Zambia.

The overall aim of this study is to document the burden of ETEC associated diarrhoea in Zambian children under 3 years of age.

DETAILED DESCRIPTION:
This study seeks to determine diarrhoea aetiology, calculate the incidence of moderate-to-severe ETEC-associated diarrhea, and describe the frequency of ETEC colonization factors and enterotoxin types in children under 3 years old in Zambia.

These data are required for the design of an anticipated phase 3 trial of the leading ETEC vaccine (ETVAX®) that will be evaluated in Zambia from 2021 onwards.

The following are the research questions that this study seeks to answer:

1. What is the incidence of MSD with confirmed ETEC aetiology in children under three years old in Zambia?
2. What are the prevalent colonization toxins and factors (CFs) in diarrhoeagenic isolates of ETEC infections in children in Zambia?
3. What are the other common pathogens causing diarrhoea in Zambian children?

This prospective, observational, longitudinal study is proposed at five health facilities in Lusaka. The proposed study sites are Chawama, George, Kanyama, Chainda, and Matero Health Facilities. These facilities are located within typical peri-urban settlements of Lusaka and serves communities with a cumulative total population of over 1 million people. The study will be done in two stages beginning with a household census in the study catchment area of the participating health facilities and then followed by the passive diarrhoea surveillance stage. A surveillance system for passive case detection of diarrhoea will be set up at each facility for the 12-months of the project to detect any seasonal variations of disease burden. Prior to commencement, several community sensitization activities will be conducted within the catchment areas of the health facility.

A stool sample will be collected from each participant who presents to the health facility and is eligible for enrollment. All research samples will be collected at the study site and laboratory assays will be performed as per written SOPs and will be a part of the study documentation. All the samples will be processed in Zambia using the Novodiag® platform. The Novodiag® (Mobidiag Ltd, Finland) is a novel multiplex molecular platform that is based on real-time PCR and microarray technology and can identify various gastroenteritis causing bacteria, parasites and viruses as well as carry out antimicrobial resistance gene testing of organisms.

ELIGIBILITY:
Inclusion Criteria:

* A child < 36 months old at the time of enrolment.
* A child presenting with diarrhoea (i.e. > 3 episodes of looser than normal stools in 24 hours) at a health facility within the study catchment area and in possession of a study ID number.
* Parents of eligible children, able to understand the study information and give informed consent by signature or thumbprint. (NB. illiterate participants will be able to give consent in the presence of an impartial witness)
* Children living within the study catchment area served by each participating health facility and in possession of a study ID number
* The parent/s who is willing to comply with all stipulated study procedures.
* Parents who are willing to allow their child to submit a stool sample for testing.

Exclusion Criteria:

* Children presenting to the health facility without a study ID number
* Any child born after the Census has taken place
* Any child currently participating in the OEV124 study

Max Age: 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: This study is a multi-site longitudinal observation study, to be conducted at Matero First Level Hospital, Chawama First Level Hospital, George Clinic, Kanyama First Level Hospital and Chainda clinic in Lusaka. The facilities are situated in a typical peri-urban settlement area of Lusaka and serves a community with a combined population of about 1 million. We assume that all sites have similar incidence of ETEC diarrhoea, therefore, each of the 5 sites will enroll 1350 children bringing our total sample size for the study to 6,750 participants.
Sampling Method: Probability Sample
Enrollment: 6828 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2021-10-15 (Actual)

PRIMARY OUTCOMES:
Incidence of MSD ETEC diarrhoea in Zambia. | 12 months
  Number of cases of moderate to severe diarrhoea (MSD) with confirmed ETEC aetiology in children under 3 years old in Zambia and the risk factors for ETEC diarrhoea

SECONDARY OUTCOMES:
Virulence factors of ETEC isolates | 12 months
  The prevalent ETEC virulence factors (LT, STh and STp ) and colonisation factors (CFA/I, CS1, CS2, CS3, CS4, CS5, CS6, CS7, CS8, CS12, CS14, CS17) in diarrhoeagenic isolates of ETEC.
The common pathogens causing MSD in children less than 3 years | 12 months
  Number of diarrhoea cases due to Shigella, campylobacter coli/jejuni, Clostridium difficile, EAEC, EHEC, EPEC, Salmonella, Vibrio cholerae, Vibrio parahaemolyticus and Yersinia enterocolitica.
Seasonality of ETEC diarrhoea | 12 months
  The incidence of ETEC positive diarrhoea cases per month for 1 year.
Antimicrobial resistance pattern of ETEC | 12 months
  AMR pattern for ETEC will be determined by presence or absence of 9 major carbapenemases genes (KPC, NDM, VIM, IMP, OXA-23, OXA-24, OXA-48/181, OXA-51, OXA-58)

CONTACTS AND LOCATIONS:
Overall Officials: Roma Chilengi, MBChB, Principal Investigator — Centre for Infectious Disease Research in Zambia; Monde Muyoyeta, MBChB, Principal Investigator — Centre for Infectious Disease Research in Zambia
Locations (4):
- Zambia (4):
  - Chawama First level hospital, Lusaka
  - George Clinic, Lusaka
  - Kanyama First Level Hospital, Lusaka
  - Matero Clinical Research Site, Chainda South CRS, Lusaka

IPD SHARING:
Plan to Share IPD: Undecided